CLINICAL TRIAL: NCT01616342
Title: Investigator Initiated Trial- Management of Chronic Pain in Military Patients With Injuries Sustained During Active Duty. Comparison of Spinal Cord Stimulation and Comprehensive Medical Management
Brief Title: Management of Chronic Pain in Military Patients With Injuries Sustained During Active Duty
Acronym: War Wounded
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sceptor Pain Foundation (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 29SEPT2011
Record Dates: First submitted 2011-10-26; First posted 2012-06-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Extremity Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comprehensive Medical Management (Active Comparator): Comprehensive Medical Management will include analgesic management in accordance with guidelines and practices at the site.
  Interventions: Device: Spinal cord stimulator
- Spinal Cord Stimulation (SCS) (Active Comparator): Subjects assigned to Arm A, CMM + SCS, will be treated with electrical pulses from a surgically implanted Precision Plus® SCS System (Boston Scientific Corporation).
  Interventions: Device: Spinal cord stimulator

INTERVENTIONS:
Device: Spinal cord stimulator — Precise (TM) spinal cord stimulator from boston scientific, and comprehensive mdedical management.

SUMMARY:
The purpose of this study is to determine the degree to which spinal cord stimulation added to comprehensive medical management can provide increased relief of chronic pain in patients with injuries sustained while on active military duty, measured by patient assessments of pain.

DETAILED DESCRIPTION:
The study population includes combat-injured patients and other patients injured while on active duty who experience chronic pain as a result of the injury and who receive treatment as active duty military personnel at Department of Defense facilities or through the Department of Veteran's Affairs. The population will include patients with pain related to limb amputation, and patients eligible for care in the Veteran's Administration Polytrauma Network program (Polytrauma Veterans) or for management of similar injuries within the Department of Defense health care system. Study subjects will have complex problems that are difficult to treat with current standard rehabilitative approaches. The circumstances of these patients' injuries create a substantial societal interest in determining and providing the best achievable rehabilitation, an interest that combines the expectation that medical science will advance the quality of medical care, practical benefits to subjects and society of returning patients to active duty or employment, and the moral imperative to support persons injured while defending our national security.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a veteran or active duty service member injured while on active military duty receiving care for pain related to the injury(ies) in the Department of Defense health care system or through the Department of Veteran's Affairs.
* Subject is 18 years of age or older.
* The elapsed time since the active-duty injury leading to chronic pain is not less than 3 months.
* Subject reports constant or daily episodes of injury-related pain of at least moderate severity, graded 4 or higher on an 11-point NPRS (point estimate by subject and Investigator at time of enrolment based on overall pain or pain at a specific site). Pain may be nociceptive, neuropathic, or mixed. Phantom pain associated with amputation of an extremity or extremities is allowed.
* Attempts to control pain with commercially available systemic analgesics have not provided adequate relief, in the judgment of the managing physician and subject.
* Subject is able to localize site(s) of pain. At least one site of daily pain contributing to moderate severity (Inclusion Criterion 4) and intractability (Inclusion Criterion 5) must be in an extremity, or phantom pain at the site of an amputated extremity. If the extremity site of pain is not an amputated limb, then the pain must have a neuropathic component. This site is identified as the site of Target Pain (TP) for efficacy evaluations during the trial.
* Subject is an acceptable candidate for surgical placement of an indwelling spinal cord stimulation device.
* Subject is judged an appropriate candidate for treatment using the available techniques and interventions encompassed within the protocol's definition of comprehensive medical management.
* For the duration of the trial, subject is willing to limit interventions for control of chronic pain to those approved by the Investigator.
* The subject is judged psychologically appropriate for either treatment intervention, based on the impression of an interviewing psychologist or psychiatrist.
* Subject provides informed consent.

Exclusion Criteria:

* Subject experiences phantom pain associated with amputation of both an upper and lower extremity.
* Subject has headache or visceral truncal pain or other non-musculoskeletal pain as the only pain that results in constant or daily scores of ≥4 on the 11-point NPRS.
* Subject has spinal disease that would, in the judgment of the investigator, - Subject has ongoing chronic infection or a medical condition associated with an unacceptably increased risk of infection related to device implantation.
* Subject has a current diagnosis or history of psychosis, cognitive impairment, hallucinations, or unexplained loss of consciousness, whether or not related to a combat injury that, in the opinion of the investigator, would exclude the patient from participating in the trial.
* Subject has a cardiac pacemaker.
* Subject has any significant medical or psychiatric condition that would interfere with the conduct of the study or with the outcome measures.
* Subject is pregnant or is breast feeding.
* Subject has participated in any drug or device trial in the past 30 days.
* Subject has any planned elective or semi-elective surgery during the 6 months of the Primary Treatment Phase, including stump revisions or grafting.
* Subject has a psychological condition of great enough severity that it would unacceptably increase the medical risks associated with implantation and care of the devices required for the treatment on the CMM + SCS arm, or would likely interfere with the subject's ability to sustain participation in a research study of long duration. Investigators are encouraged to include the medical monitor and the coordinating investigator in discussions about individual candidate subjects who have psychological diagnoses as part of the polytrauma syndrome before enrollment or treatment on this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain score | 144 weeks
  Change from Baseline to Week 24 in weekly mean of average daily pain scores at the target site of pain (target pain, TP), based on an 11-point Numerical Pain Rating Scale (NPRS), by treatment group.

SECONDARY OUTCOMES:
change in related pain | 144 weeks
  Change from Baseline to Week 24 and Week 144 in subjects' experiences related to pain, using the Pain Outcomes Questionnaire for Veterans Affairs (Intake and Discharge; POQ-VA), by treatment group.
change in mean daily pain score | 144 weeks
  Change from Baseline to Week 24 in weekly mean of average daily pain scores for overall pain (OP), based on an 11-point Numerical Pain Rating Scale (NPRS), by treatment group.
change in mean pain per treatment group | 144 weeks
  Change from Baseline to Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 36, Week 48, Week 72, Week 96, Week 120, and Week 144 in weekly mean of average daily pain scores for TP and OP, based on the 11-point NPRS, by treatment group.
change in MPQ per treatment group | 144 weeks
  Change from Baseline to Week 24, Week 48, Week 96, and Week 144 in pain evaluation, measured by the McGill Pain Questionnaire (MPQ), by treatment group.
change in spine related pain | 144 weeks
  Change from Baseline to Week 24, Week 48, Week 96, and Week 144 in spine-related pain, measured by the Modified Oswestry Pain Questionnaire, by treatment group.
change in neuropathic pain | 144 weeks
  Change from Baseline to Week 24, Week 48, Week 96, and Week 144 in neuropathic pain, measured by the Neuropathic Pain Scale (NPS), by treatment group
analgesic efficacy | 144 weeks
  Overall analgesic efficacy, measured by Investigator and Subject using categorical global scores of change at Week 24 and Week 144 (GIC-I, GIC-S), by treatment group.
pain relief using a categorical scale | 144 weeks
  Assessment of pain relief, measured by the Subject using a categorical 5-point scale (None =0, A Little =1, Some =2, A Lot =3, or Complete =4) at Week 24 and Week 144, by treatment group
change in mood | 144 weeks
  Change from Baseline to Week 24, Week 48, Week 96, and Week 144 in patient mood, measured by the Profile of Mood Survey (POMS), by treatment group.
change in emotional status | 144 weeks
  Change from Baseline to Week 24, Week 48, Week 72, and Week 144 in patient emotional status (mood), measured by the Beck Depression
change in anxiety | 144 weeks
  Change from Baseline to Week 24, Week 48, Week 72, and Week 144 in patient anxiety, measured by the Impact of Events - Revised (IES-R) scale and by the Post Traumatic Stress Disorder Checklist (PCL), by treatment group.
change in quality of life | 144 weeks
  Change from Baseline to Week 24, Week 48, Week 96, and Week 144 in quality of life, measured by the SF-36 Health Survey, by treatment group.
effectiveness of intervention | 144 weeks
  Overall effectiveness of intervention as measured by number (%) of subjects who withdraw prior to Week 24, prior to Week 48, prior to Week 96, and prior to Week 144, due to lack of efficacy.
Functional effectiveness of intervention | 144 weeks
  Functional effectiveness of intervention as measured by number (%) of subjects who return to duty (active duty subjects) or return to employment (subjects treated as veterans) at Week 24, Week 48, Week 96, and Week 144.
Functional effectiveness of interventions via activity scores | 144 weeks
  Functional effectiveness of interventions as measured by daily mean and peak activity scores and numbers of days with sedentary or moderate activity levels based on data downloads from the 3-D accelerometer at Baseline, during the 2-week interval prior to Week 12, and for the 2-week intervals preceding visits at Week 24, Week 48, Week 96, and Week 144.
change in sleep | 144 weeks
  Change in Chronic Pain Sleep Inventory (CPSI), Baseline to Week 24, Week 48, Week 96, and Week 144, by treatment group.
urine drug tests | Baseline, week 6, week 12, week 24
  Number (percentage) and change from Baseline in number (percentage) of subjects with non-adherence to the prescribed analgesic drug regimen (detection of non-prescribed medication/metabolite or non-detection of prescribed medication/metabolite) on urine drug tests (UDT), at Baseline, Week 6, Week 12, and Week 24.
Effect of demographic characteristics | 144 weeks
  Effect of demographic characteristics, combat exposure (measured by the combat exposure scale administered at Baseline), elapsed time since injury, site of injury, and type of injury (blast injury, penetrating wound, burn, amputation, combat versus non-combat, other) on the effectiveness of intervention measured by the subject reports of pain and pain relief, overall effectiveness scores, and efficacy scales, by treatment group.
predictive value of the change in NPRS average pain scores | Week 24, Week 48, Week 96, and Week 144
  For subjects assigned to Arm A (CMM + SCS), the predictive value of the change in NPRS average pain scores (both TP and OP) from Baseline to the pre-implantation trial week for the scores observed at Week 24, Week 48, Week 96, and Week 144.
Analgesic benefit | 144 weeks
  Analgesic benefit of crossover to the non-assigned treatment arm, measured in subjects who change from the assigned arm to the alternative arm before Week 24, using the efficacy assessments recorded prior to crossover (removal or implantation of the SCS device), summarized as LOCF values at Week 24, with efficacy assessments during the weeks following the crossover event, counted as if the crossover event initiated (re-started) the Primary Treatment Phase.
Safety and tolerability of analgesic interventions | 144 weeks
  Safety and tolerability of analgesic interventions, measured by spontaneously reported adverse events, serious adverse events, and adverse events leading to early withdrawal, by treatment group.
Tolerability of analgesic interventions | 144 weeks
  Tolerability of analgesic interventions as measured by total number of hospital days experienced by the subject, including hospital days required for study-related interventions and hospital days resulting from adverse events and in-patient management of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rauck, MD, Principal Investigator — The Center for Clinical Research; Derry Ridgeway, MD, Study Chair — SRA International
Locations (1):
- Center for Clinical Research, Winston-Salem, North Carolina, United States